CLINICAL TRIAL: NCT05325749
Title: Development of the Technology and Methodology for Generation of the Genetic Passport (Genetic Health Record) of Newborn and Application Thereof to Estimate the Mid and Low Penetrance Hereditary Disorders Frequencies in Russian Population and to Uncover Genetic Factors Determining Severe Monogenic Conditions
Brief Title: Whole Exome Screening of Newborns
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federal State Budget Institution Research Center for Obstetrics, Gynecology and Perinatology Ministry of Healthcare (Other Government)
Responsible Party: Sponsor
Other Study IDs: Examen
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2021-12

CONDITIONS: Infant, Newborn
Keywords: newborn; whole exome; genetic screening
MeSH Terms: interventions — Mass Screening; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- unaffected: newborns without developmental features having no variations according to an inherited diseases screening;
  Interventions: Genetic: Screening; Genetic: Family history record; Other: Questionnaire survey
- affected: newborns showing either phenotypic features or deviations according to MS screening
  Interventions: Genetic: Screening; Genetic: Family history record; Other: Questionnaire survey; Genetic: Diagnostic
- refused families: parents refused to enroll their newborns to the study
  Interventions: Other: Questionnaire survey
- unaffected born prematurely: newborns without specific developmental features having no variations according to an inherited diseases screening, born before term
  Interventions: Genetic: Screening; Genetic: Family history record; Other: Questionnaire survey; Genetic: Selective screening
- unaffected wirh family history: newborns without developmental features having no variations according to an inherited diseases screening but with affected relative(s)
  Interventions: Genetic: Screening; Genetic: Family history record; Other: Questionnaire survey; Genetic: Selective screening
- unaffected wirh prenatal phenotype: newborns without developmental features at birth and on, having no variations according to an inherited diseases screening which had been observed to show signs of developmental features during prenatal ultrasound examination
  Interventions: Genetic: Screening; Genetic: Family history record; Other: Questionnaire survey; Genetic: Selective screening

INTERVENTIONS:
Genetic: Screening — Whole exome sequencing will be done and all infants will receive a report which will include pathogenic or likely pathogenic variants identified in genes associated with childhood-onset diseases for which specific care or prevention protocols are available. Families signed additional informed consent will receive an advanced report including variants with no care or prevention available, mid or low risk variants, and variants with late onset or those suggesting relatives to undergo screening.
  Groups: affected; unaffected; unaffected born prematurely; unaffected wirh family history; unaffected wirh prenatal phenotype
Genetic: Family history record — Families enrolled to the study will receive a genetic consult during which a family history will be taken concerning the inherited conditions.
  Groups: affected; unaffected; unaffected born prematurely; unaffected wirh family history; unaffected wirh prenatal phenotype
Other: Questionnaire survey — Families invited to the study will be asked to undergo a questionnaire survey regarding the reasons to accept or refuse the study, the familiarity of the aims, methods and outcomes of the study as well as the satisfaction.
Genetic: Diagnostic — The results of whole exome sequencing will be analysed according to the infant's phenotype in addition the the general screening pipeline
  Groups: affected
Genetic: Selective screening — The results of whole exome sequencing will be analysed according to the data of prenatal ultrasound examination, family history and other available alarming information in addition the the general screening pipeline
  Groups: unaffected born prematurely; unaffected wirh family history; unaffected wirh prenatal phenotype

SUMMARY:
The aim of the study is to obtain the initial experience of the inclusive genetic screening of newborn.

Two groups of newborns born in RCOGP will be enlisted to the study:

1. newborns without developmental features having no variations according to an inherited diseases screening;
2. newborns showing either phenotypic features or deviations according to MS screening.

The residual volume of the cord blood of all newborns form both groups will be collected and subjected to the whole exome sequencing. The sequencing data will be analyzed in "screening" mode for the first group while for the second group analysis will be performed taking the respective phenotype into account.

The study is planned to cover 7000 newborns in total.

ELIGIBILITY:
Group 1 (newborns without features):

Inclusion Criteria:

* Infants born in the RCOGP, showing no development features and with no inherited diseases revealed by common screening
* Informed consent signed by a newborn's representative

Exclusion Criteria:

* Parents refuse to participate
* Parent(s) younger 18 years
* Parent(s) unable to make decisions
* The infant is older 30 d
* Blood cannot be collected from the infant

Group 2 (newborns with phenotypic features)

Inclusion Criteria:

* Infants showing either phenotypic features or deviations according to MS screening
* Informed consent signed by a newborn's representative

Exclusion Criteria:

* Parents refuse to participate
* Parent(s) younger 18 years
* Parent(s) unable to make decisions
* Blood cannot be collected from the infant
* Detailed description of the phenotype is not available
* The infant's exome has been already sequenced

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All infants born in the RCOGP or under treatment in an ICU departmetn of the RCOGP
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2021-07-10 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Estimate the frequency of revealing patients carrying genotype associated with a monogenic disese. | 3-5 months
  The manifestation of pathogenic or likely pathogenic variants leading to a monogenic disease presenting during early age.
  A genotype is considered having risk of developping a monogenic disease in case pathogenic or probably pathogenic variants are detected corresponding to the inheritance model.
Phenotype-associated variants | 2 weeks - 2 months
  Pathogenic, likely pathogenic variants or variants of uncertain significance corresponding to the observed clinical conditions
Motivations for refuse to participate | 1 day
  Questionnaire answers provided by families refused to enroll
Acceptance of advanced screening | 1 day
  Questionnaire answers provided by families accepted screening for variants of low penetrance, no care available etc.

SECONDARY OUTCOMES:
Oncological risk | 1 day
  Pathogenic or a likely pathogenic variant causing high risk of developping a cancer
Cardiological risk | 1 day
  Pathogenic or a likely pathogenic variant causing high risk of developping a cardiomyopathy or a sudden cardiac death
Recessive carriers | 1 day
  Inheritance of a pathogenic or a likely pathogenic variant causing to an autosomal recessive disease

CONTACTS AND LOCATIONS:
Overall Officials: Dmitriy Y Trofimov, DSc, Study Director — Federal State Budget Institution Research Center for Obstetrics, Gynecology and Perinatology Ministry of Healthcare
Locations (1):
- Federal State Budget Institution Research Center for Obstetrics, Gynecology and Perinatology Ministry of Healthcare, Moscow, Russia

REFERENCES:
- [Derived] Kochetkova TO, Maslennikov DN, Tolmacheva ER, Shubina J, Bolshakova AS, Suvorova DI, Degtyareva AV, Orlovskaya IV, Kuznetsova MV, Rachkova AA, Sukhikh GT, Rebrikov DV, Trofimov DY. De Novo Variant in the KCNJ9 Gene as a Possible Cause of Neonatal Seizures. Genes (Basel). 2023 Jan 31;14(2):366. doi: 10.3390/genes14020366. PMID 36833293